CLINICAL TRIAL: NCT06846177
Title: Effects Of Graded Activity Training and Task-Oriented Training on Fatigue in Post-Stroke Patients
Brief Title: Graded Activity Training and Task- Oriented Training on Post-Stroke Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sahar Khalid
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Post-Stroke Fatigue
Keywords: Task oriented training; Graded activity training; Post stroke; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Activity Training (Experimental): Graded Activity Training
  Interventions: Other: Graded Activity Training
- Task Oriented Training (Active Comparator): Task Oriented Training
  Interventions: Other: Task-Oriented Training

INTERVENTIONS:
Other: Graded Activity Training — 4 types of progressive activities of 2 hour session two times/week with resting periods of 30 mins. Activities consist of treadmill walk ,walk on floor, core muscles exercises ,home tasks .
  To ensure the proper heart rate and loads during the exercises, measurements of individual heart rate and muscle strength are taken during the first session (baseline) with HR Tracking portable device and also during the session to continuously monitor HR of the Patient. To withdraw or adjust the training intensity for each patient Borg's Scale of Perceived Exertion is used throughout the session for monitoring Training intensity of endurance, muscle training, individual's effort and exertion level.
  Arms: Graded Activity Training
Other: Task-Oriented Training — 4 task oriented physical fitness activities which include walk on floor, walk on inclined surface using treadmill ,sit to stand , stair climbing and descending for duration of 2 hour session with frequent breaks. Each treatment session began with 10 minutes of warm-up exercise, which consisted of passive stretching of the calf muscles, hamstring, and hip adductors. The level of difficulty and frequency for each task were gradually increased during the 6 weeks with the patients consent.10 minutes of cool down at the end of each treatment session.
  Arms: Task Oriented Training

SUMMARY:
The aim of this randomized controlled trial is to determine the effects of Graded Activity Training and Task Oriented Training on Fatigue in Post-Stroke Patients. Until now there is very limited work found on fatigue so this will increase quality of life in stroke patients and potentially reduce burden on healthcare system.

DETAILED DESCRIPTION:
Post stroke fatigue (PSF) is one of the most common outcomes of stroke. PSF is defined as "overwhelming feeling of exhaustion or tiredness" as a result of stroke PSF is an undesirable outcome by which patient's ability in study participation, adherence to medication and effectiveness of rehabilitation decrease which is unrelated to exertion, and does not typically improve with rest. Prevalence rate of PSF ranges between 25% and 85% One out of two stroke survivors experience post-stroke fatigue. The relationship between physical deconditioning and fatigue is bidirectional there was a negative relationship between fatigue and aerobic fitness in chronic stroke. PSF may arise from physical deconditioning (physical fatigue). Therefore, improving physical endurance through physical activity training could potentially reduce fatigue complaints.

The rationale of this study is to determine how task-oriented training and graded activity training effect stroke patient's levels of fatigue and to develop an improved fatigue management intervention protocol. This study will also determine effects of how both interventions affect Mobility and Gait. By doing so, we can identify a more effective PSF intervention plan, which will help reduce the burden on the healthcare system and will lessen strain on caregivers and in turn enhance patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female of age 40 to 60 years.
* Patient with both ischemic or hemorrhagic stroke.
* Patient with both right and left hemiplegia.
* Checklist Individual (CIS-F) fatigue score of 40 or more.
* Patients who had sustained a stroke more than 4 months before recruitment.
* Patients who can independently walk for 10 meters (about 33 feets)

Exclusion Criteria:

* Patients with severe comorbid health conditions (such as cardiac diseases, pulmonary diseases like COPD, Orthopedic Conditions Arthritis, joint replacements).
* Patients with uncontrolled diabetes, hypertension, Depression and Anxiety.
* Patients who are not willing to participate.
* Patient with any medications that can affect their ability to engage in physical training program like Antidepressants, Beta-Blockers, corticosteroids etc.
* Pregnant women.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Fatigue Assessment scale (FAS) | 6 weeks
  The FAS is a 10-item scale is used to evaluate symptoms of chronic fatigue. In contrast to other similar measures description of the fatigue experienced is presented for the total score of l<22 indicates normal, levels of fatigue between 22 to 34 indicates mild to moderate fatigue and score 35 or more indicates severe fatigue

SECONDARY OUTCOMES:
Timed Up and go test(Mobility) | 6 weeks
  The Timed Up and Go (TUG) is a commonly used outcome measure that is used to assess mobility and fall risk among older adults. It is a simple test that measures how quickly you can stand up, walk 10 feet, turn around, walk back, and sit down. cut off score of ≥12 seconds indicates high risk of fall.
Dynamic gait index (Gait) | 6 weeks
  The DGI is 8 item scale to assess gait. The scoring of the DGI is based on a 4 point scale ranging from 0 to 3, with 0 indicating severe impairment and 3 indicating normal ability. The best performance total score is 24. A low composite DGI score thus indicates greater impairment

OTHER OUTCOMES:
Checklist individual strength-Fatigue (CIS-F) (Screening tool) | 1st week
  a 20-items questionnaire for fatigue and is used in various illnesses, including Myalgic encephalomyelitis/chronic fatigue syndrome CSF.
  4 components in the remaining 20 questions. These were easy to interpret and were called Subjective Fatigue 8 items, Concentration 5 items, Motivation 4 items, Physical activity 3 items. A higher score indicates more fatigue. cutt off score 40 or above will be selected for inclusion criteria
Borg's Rating of Perceived Exertion (Monitoring Tool | 6 weeks
  The Borg Rating of Perceived Exertion (RPE) scale is a tool for measuring an individual's effort and exertion, breathlessness and fatigue during physical work .The Borg RPE scale rates exertion from a scale of 6 (no exertion) to 20 (maximum effort). A rating between 12 to 14 typically reflects a moderate or somewhat hard level of intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Aroosa Tariq, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute of Rehabilitation Sciences, Mansehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No